CLINICAL TRIAL: NCT01476358
Title: A Randomized Controlled Trial in Human Neonates to Determine the Effect of Vitamin A Supplementation on Immune Responses
Brief Title: Effect of Vitamin A Supplementation on Immune Responses in Human Neonates
Acronym: NNVAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: RPC389
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Vitamin A Deficiency
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Vitamin A; retinol palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin A (Active Comparator): Capsule containing oil vehicle with Vitamin A (retinyl palmitate). Capsules are prepared by the manufacturer (Strides Arcolab Limited, India) and assigned blinded codes by World Health Organization officials.
  Interventions: Dietary Supplement: Vitamin A (retinyl palmitate).
- Placebo (Placebo Comparator): Capsule containing oil vehicle withOUT Vitamin A (retinyl palmitate). Capsules are prepared by the manufacturer (Strides Arcolab Limited, India) and assigned blinded codes by World Health Organization officials.
  Interventions: Dietary Supplement: Vitamin A (retinyl palmitate).

INTERVENTIONS:
Dietary Supplement: Vitamin A (retinyl palmitate). — Active Comparator (Vitamin A): 1 capsule containing oil carrier and 50,000IU Vitamin A, within 48hs of birth
  Placebo Comparator: 1 capsule containing oil carrier and 0IU Vitamin A, within 48hs of birth

SUMMARY:
Vitamin A supplementation (VAS) significantly reduces all-cause mortality when given after 6 months of age, but has a null or detrimental effect when given between 1-5 months. Studies of neonatal VAS (NNVAS) have produced conflicting findings. These age-pattern variations might result from immunological interactions between VAS and vaccines. The potential efficacy of NNVAS is being retested in 3 large new intervention trials with mortality as endpoint. Complementary mechanistic studies in animals and in human infants in The Gambia (this proposal) and Bangladesh have been commissioned to run in parallel.

The investigators will use a 2-arm double blind RCT to test whether NNVAS modulates the early ontogeny of human immune development. Neonates, recruited through a peri-urban clinic in The Gambia, will receive either 50,000 International Units (IU) VAS orally within 48 hours of birth (intervention group, n=100) or a placebo (control group, n=100). Male and female neonates will be randomized separately at enrolment for later analyses by sex. All infants will be followed up from birth to age 1 year. A broad panel of immunological outcomes will examine whether NNVAS: a). normalises thymic development (thymic index by ultrasound); b). skews mycobacterial and recall antigen responses towards a Th2 profile; c). diminishes Th1 and Th17 reactivity to mycobacterial and recall antigens; d). diminishes the tuberculin skin test (TST) response; e). causes increased innate immune reactivity; f). increases the frequency of circulating regulatory T cells (Tregs) expressing gut homing receptors; g). enhances B cell immune responses after routine vaccination (increase of B cell numbers and activation status); h). increases circulating IgA in mucosal immune compartment, especially oral polio vaccine (OPV) specific IgA post-vaccination; i). decreases bacterial translocation, by improving mucosal barrier function; and j). decreases markers of infection or inflammation. Growth and morbidity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* singleton birth,
* birth weight ≥1,500g,
* mother over 18 years willing to participate and residency within the study area.
* Birth vaccinations and vitamin A supplement must be administered within 48 hours of birth.

Exclusion Criteria:

* Infants having a congenital disease,
* a serious infection at birth
* an inability to feed (initially assessed by the lack of the suck reflex),
* mothers who are seriously ill at time of enrolment (defined as bed bound for more than 24 hours),
* mother participating in other studies,
* mothers who are HIV positive.

Ages: 5 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of circulating Tregs expressing gut homing receptors in infant participants. | 17 week post-supplementation

SECONDARY OUTCOMES:
Difference in Thymus size in infant participants | 1, 6, 12 and 17 weeks
  Assessed by ultrasonic analysis.
Difference in B cell immune responses after routine vaccination in infant participants | 6 and 17 weeks
  Assessed as an increase in B cell numbers and activation status.
Improved mucosal barrier function in infant participants | 6 and 17 weeks
  Assessed by quantifying bacterial translocation into the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna LR McDonald, BSc (Hons) MSc PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Medical Research Council, The Gambia Unit, Fajara, The Gambia

REFERENCES:
- [Derived] McDonald SL, Savy M, Fulford AJ, Kendall L, Flanagan KL, Prentice AM. A double blind randomized controlled trial in neonates to determine the effect of vitamin A supplementation on immune responses: The Gambia protocol. BMC Pediatr. 2014 Apr 4;14:92. doi: 10.1186/1471-2431-14-92. PMID 24708735